CLINICAL TRIAL: NCT00208312
Title: A Phase III, Randomized, Double-Blind Study of Intravenous CVT-3146 Versus Adenoscan® in Patients Undergoing Stress Myocardial Perfusion Imaging
Brief Title: ADVANCE MPI 2: Study of Regadenoson Versus Adenoscan® in Patients Undergoing Myocardial Perfusion Imaging (MPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Philip Sager, Vice President, Clinical Research, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CVT 5132
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease
Keywords: Lexiscan; Regadenoson; Adenoscan®; Adenosine; SPECT Myocardial Perfusion Imaging; Reversible Perfusion Defect
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson; Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Regadenoson
  Interventions: Drug: Regadenoson
- 2 (Active Comparator): Adenoscan
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Regadenoson — 0.4 mg, bolus intravenous injection
  Other Names: Lexiscan; CVT-3146
  Arms: 1
Drug: Adenosine — 0.14 mg/kg/min for 6 minutes, intravenous infusion
  Other Names: Adenoscan
  Arms: 2

SUMMARY:
Adenoscan® (adenosine) is an approved pharmacological stress agent indicated as an adjunct to thallium-201 myocardial perfusion scintigraphy in patients unable to exercise adequately. The investigational drug, regadenoson (CVT-3146) is a selective A2A adenosine receptor agonist, the receptor responsible for coronary vasodilation, and is being studied for potential use as a pharmacologic stress agent in myocardial perfusion imaging (MPI) studies. This study will compare the safety and efficacy of regadenoson to that of Adenoscan in detecting reversible myocardial perfusion defects.

DETAILED DESCRIPTION:
ADVANCE MPI 2 is a multi-national, double-blind, randomized, active-controlled, parallel group clinical trial to evaluate the safety and efficacy of regadenoson in SPECT MPI compared to that of the approved pharmacological stress agent, Adenoscan. Patients referred for a clinically indicated pharmacological stress MPI study will be eligible for enrollment. The trial is designed: (1) to compare the pharmacological stress SPECT images obtained with regadenoson to those obtained with Adenoscan, and (2) to compare the safety and tolerability of the two stress agents.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a clinically indicated pharmacological stress SPECT myocardial perfusion imaging study

Exclusion Criteria:

* Any condition precluding the safe administration of Adenoscan for a SPECT myocardial perfusion imaging study
* Pregnant or breast-feeding, or (if pre-menopausal), not practicing acceptable method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of regadenoson to Adenoscan for use in SPECT myocardial perfusion imaging in assessing reversible perfusion defects | After radiopharmaceutical administration

SECONDARY OUTCOMES:
Safety and tolerability comparison of regadenoson to Adenoscan | Up to two weeks
Additional comparisons of images obtained with regadenoson to those obtained with Adenoscan | After radiopharmaceutical administration

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple study locations (see Central Contact); CV Therapeutics, Inc., Palo Alto, California, United States

REFERENCES:
- [Result] Iskandrian AE, Bateman TM, Belardinelli L, Blackburn B, Cerqueira MD, Hendel RC, Lieu H, Mahmarian JJ, Olmsted A, Underwood SR, Vitola J, Wang W; ADVANCE MPI Investigators. Adenosine versus regadenoson comparative evaluation in myocardial perfusion imaging: results of the ADVANCE phase 3 multicenter international trial. J Nucl Cardiol. 2007 Sep-Oct;14(5):645-58. doi: 10.1016/j.nuclcard.2007.06.114. PMID 17826318
- See also: Adenoscan® — http://www.adenoscan.com